CLINICAL TRIAL: NCT04502641
Title: A Randomized Phase III Comparing Sequential Therapy With Induction Chemotherapy/Chemoradiation To Cisplatinum-Based Chemoradiotherapy in Locally Advanced Hypopharyngeal Carcinoma
Brief Title: Induction Chemotherapy in Locally Advanced Hypopharyngeal Carcinoma: a Randomised Phase 3 Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Zhen-Wei Peng, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: hypopharyngeal SCC 001
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Hypopharyngeal Cancer
Keywords: hypopharyngeal carcinoma; chemotherapy; radiotherapy; prognosis
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — Docetaxel; Paclitaxel; Fluorouracil; Cisplatin; Radiotherapy, Intensity-Modulated; Platinum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (Experimental): Patients receive induction chemotherapy with docetaxel-based, with or without cisplatin or fluorouracil. Treatment repeats every 21 days for 3 courses. Then, patients receive cisplatin on day 1 day 21, 3 weeks as one cycle and undergo concurrent radiotherapy once daily, 5 days a week, for 6 to 7 weeks.
  Interventions: Drug: Docetaxel; Drug: 5-fluorouracil; Drug: Cisplatin; Radiation: Intensity Modulated Radiation Therapy; Drug: Platinum
- Arm II (Active Comparator): Patients receive cisplatin on day 1 day 21, 3 weeks as one cycle and undergo concurrent radiotherapy once daily, 5 days a week, for 6 to 7 weeks.
  Interventions: Radiation: Intensity Modulated Radiation Therapy; Drug: Platinum

INTERVENTIONS:
Drug: Docetaxel — 60mg/m2 on day 1, 3 weeks as one cycle, for 3 cycles.
  Other Names: Taxol
  Arms: Arm I
Drug: 5-fluorouracil — 600 mg/m² per day as a continuous 120 h infusion on days 1-5, 3 weeks as one cycle, for 3 cycles.
  Arms: Arm I
Drug: Cisplatin — 60mg/m2 on day 1, 3 weeks as one cycle, for 3 cycles.
  Arms: Arm I
Radiation: Intensity Modulated Radiation Therapy — The treatment consisted of definitive radiotherapy with conventional fractionation, a total dose of 68-70 Gy to PTVp, 62-68 Gy to PTVn, 60-62 Gy to PTV-HR, and 50-54 Gy to PTV-LR.
Drug: Platinum — 100mg/m2 on day 1, 3 weeks as one cycle, during radiotherapy.

SUMMARY:
Hypopharyngeal cancer is an important part of head and neck cancer, with more than 80,000 new cases in 2018. And it is a highly aggressive cancer often diagnosed at an advanced stage. which expresses poor survival, the 5-year overall survival (OS) is about only 30%-35%. Given the complexity of these tumors, their surrounding structures, the frequent comorbidities, and the improvement of patients' requirements for quality of life, a multidisciplinary treatment approach should be applied to achieve the best oncological outcomes and to improve functional results. This benefi t of induction chemotherapy has been recorded in patients with both resectable and unresectable disease. It has also been observed in patients with laryngeal cancer treated for organ preservation. However, whether the addition of induction chemotherapy to chemoradiotherapy improves efficacy compared with chemoradiotherapy alone is unclear in hypopharyngeal cancer.We tried to observe the clinical treatment efficiency, toxic and side effects, progression-free survival time, overall survival time and quality of life of anlotinib in the treatment of patients with refractory head and neck carcinoma. Provide patients with a more optimal treatment plan and improve survival.

DETAILED DESCRIPTION:
We will prospectively collect 160 patients who were randomly assigned (in a 1:1 ratio) to receive either induction chemotherapy followed by concurrent chemoradiotherapy (group A) or definitive concurrent chemoradiotherapy (group B). Data will be stored in a private database. The process of data collection will be supervised and regular data examination will be performed.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male or female, aged 18 to 75 years; 2. Performance status (PS) score ≤ 2 points; 3. The expected survival period is more than 3 months; 4. Patients have histopathologically confirmed hypopharyngeal squamous cell carcinoma, including the piriform fossa, postcricoid region, and posterior pharyngeal wall with stage III and IVA-B (TNM stageT1-2N1-3M0/T3-4aN0-3M0) according to the AJCC 8th edition; 5. With measurable lesions: According to the evaluation criteria for the efficacy of solid tumors (Response Evaluation Criteria In Solid Tumors 1.1), the patient has at least one measurable lesion. The measurable lesion should not have received local treatment such as radiotherapy (target lesion located in the previous radiotherapy area, if it is confirmed that significant progress has occurred , And comply with evaluation standard, can also be used as target lesions); 6. No previous anti-tumor therapy, including anti-angiogenesis therapy, such as pazopanib, sunitinib, sorafenib, regorafenib, etc.; 7. Sufficient liver function: total bilirubin ≤ upper limit of normal value (ULN); glutamic oxalacetic transaminase (AST) and glutamic-pyruvic transaminase (ALT) ≤ 2 times upper limit of normal value (ULN); alkaline phosphatase ≤ 5 times upper limit of normal value (ULN); 8. Adequate renal function: creatinine clearance rate ≥80 mL/min; 9. Adequate blood function: absolute neutrophil count (ANC) ≥2×109/L, platelet count ≥100×109/L and hemoglobin ≥9g/dL; 10. No serious heart, lung and other important organ dysfunction; 11. Women of childbearing age must have taken reliable contraceptive measures; pregnancy tests (serum or urine) are negative within 7 days before enrollment, and must be non-lactating patients; and are willing to adopt appropriate during the test and within 6 months after the last treatment Methods of contraception. For men, it is necessary to agree to use appropriate methods of contraception or surgical sterilization during the trial and 8 weeks after the last dose; 12. The subjects voluntarily joined the study and signed an informed consent form with good compliance and cooperated with the follow-up.

Exclusion Criteria:

* 1. Have a history of other cancers in the past five years, radical or untreated prostate cancer (Gleason score ≤ 6), or complete treatment of breast ductal carcinoma in situ, except for patients with cured skin basal cell carcinoma or squamous cell skin cancer; 2. Patients with target lesions who have received radiation therapy or surgery (except biopsy); 3. Treatment with palliative intent; 4. A history of previous radiotherapy, chemotherapy, or surgery (except diagnostic) to the primary tumor or nodes; 5. Any severe coexisting disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (RFS) | 3 month
  Measured from the date of treatment end to recurrent/residual tumor was diagnose or to the time of the last follow-up, whichever occurred first，by means of computed tomography (CT) or magnetic resonance imaging (MRI) at each follow-up.

SECONDARY OUTCOMES:
Overall-survival (OS) | 3 month
  Defined as the interval between the time of treatment end to death or to the last date of follow-up，by means of computed tomography (CT) or magnetic resonance imaging (MRI) at each follow-up.
Adverse events rate | One month
  Adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chen, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China